CLINICAL TRIAL: NCT03046836
Title: Effects of Oxytocin on Alcohol Craving and Intimate Partner Aggression
Brief Title: Oxytocin, Alcohol Craving, and Intimate Partner Aggression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Julianne Flanagan, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54689
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Use
Keywords: Couples; Oxytocin; Aggression; Alcohol
MeSH Terms: conditions — Alcohol Drinking; Aggression | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Each participant will self-administer 40 international units (IU) intranasal Oxytocin
  Interventions: Drug: Oxytocin
- Control (Placebo Comparator): Each participant will self-administer matching saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40 IU oxytocin nasal spray
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Placebo — Saline
  Arms: Control

SUMMARY:
Alcohol use disorders (AUD) and intimate partner aggression (IPA) frequently co-occur. There are significant health and economic burdens associated with AUD and co-occurring IPA, and little empirical data to guide treatment efforts. The neuropeptide oxytocin may help mitigate both AUD and IPA. However, clinical data examining oxytocin's effects on human aggression is scant. The proposed study is designed to address these gaps in the literature by utilizing a human laboratory paradigm to test the effects of oxytocin on craving and aggression among couples with AUD and co-occurring IPA.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria indicate that participants must
* aged 18 or over
* fluent in English
* endorse at least one instance of mild or moderate physical IPA with their partner in the past 6 months as defined by the Revised Conflict Tactics Scale (CTS-2)
* both partners must be willing to participate
* one or both partners must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for an alcohol use disorder (AUD). Concurrent substance use disorders (e.g., marijuana) is acceptable provided alcohol is the participant's primary substance of choice.

Exclusion Criteria:

* Exclusion criteria include
* pregnancy or breastfeeding
* current or history of psychiatric or medical condition that could interfere with neuroendocrine function (e.g., hematological, endocrine, renal, or pulmonary disease; synthetic glucocorticoid or exogenous steroid therapy; psychotic, bipolar, eating disorders)
* Body Max Index (BMI) ≥ 39
* current suicidal ideation and intent
* severe physical or sexual IPA in the past six months as defined by the Conflict Tactics Scale (CTS-2)
* initiation of psychotropic medication in the past 4 weeks
* acute alcohol withdrawal as indicated by a score of 8 or greater on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-Ar).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julianne C Flanagan, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forkus SR, Baer MM, Giff ST, Hall E, Miles SR, Flanagan JC. The role of cognitive emotion regulation strategies on posttraumatic stress symptoms and alcohol use problems among individuals experiencing intimate partner violence. Psychol Trauma. 2025 Oct 23. doi: 10.1037/tra0002057. Online ahead of print. PMID 41129363
- [Derived] Flanagan JC, Nietert PJ, McCrady BS, Sellers S, Yates-Johnson A, Giff ST, Forkus SR. Results of a Randomized Controlled Trial Examining the Efficacy of Intranasal Oxytocin to Enhance Alcohol Behavioral Couple Therapy. J Clin Psychiatry. 2025 May 12;86(2):24m15627. doi: 10.4088/JCP.24m15627. PMID 40392716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from July 2017 through April 2021. Participants were recruited from local clinics, by using social media advertisements, and from the investigator's previous trials.
Pre-assignment Details: One hundred couples (N = 200 individuals) were enrolled using 1:1 randomization. Both partners within a couple were assigned to the same condition (oxytocin or placebo). Inclusion criteria indicated that one or both partners in each couple met DSM-5 criteria for current AUD and endorsed physical intimate partner aggression (IPA i.e., hitting, slapping) that occurred at any point during their current relationship, as assessed by the Revised Conflict Tactics Scale.
Groups:
- Oxytocin: Each participant will self-administer 40 IU intranasal Oxytocin
  Oxytocin: 40 IU oxytocin nasal spray
Period: Overall Study
Arm/Group | Oxytocin | Control
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Control | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (11.5) | 34.6 (11) | 35.4 (113)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 47 | 47 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 91 | 93 | 184
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 19 | 44
  White | 64 | 74 | 138
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 1 | 1 | 2
Relationship Status [Count of Participants; unit: Participants]
  Cohabitating | 47 | 43 | 90
  Married | 39 | 32 | 71
  Dating | 7 | 15 | 22
  Single | 2 | 4 | 6
  Separated | 1 | 2 | 3
  Divorced | 1 | 2 | 3
  Missing | 3 | 2 | 5
Alcohol Use Disorder (AUD) [Count of Participants; unit: Participants]
  Mild | 30 | 20 | 50
  Moderate | 14 | 19 | 33
  Severe | 37 | 37 | 74
  No AUD | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Craving
Description: Change in subjective alcohol craving as measured by a Visual Analogue Scale (VAS) between time point 3 (before the alcohol cue) and 4 (after the alcohol cue).
  Participants completed the VAS at 8 timepoints:
  Minute 0 (pre-OT/placebo) (Time 1) Minute 5 (pre-OT/placebo) (Time 2) OT/placebo administered at minute 10 Minute 40 (Time 3) Minute 45 - alcohol cue paradigm began Time 4 (immediately after alcohol cue) Minute 65 - TAP began Time 5 (immediately after TAP began) Time 6 (15 minutes after TAP) Time 7 (30 minutes after TAP) Time 8 (60 minutes after TAP)
  This 100mm Visual Analogue Scale (VAS) was anchored on a 100mm Likert-type scale from 0 (not at all/no craving) to 10 (extremely/maximum carving). The scale is set to 100mm in length, and the lowest value is a 0 (zero), representing no craving and and highest value is a 10 (ten) representing extreme craving.
Time Frame: Participants completed the VAS at 8 timepoints. Outcome measure represents the change in VAS scores between time point 3 (before the alcohol cue) and 4 (after the alcohol cue).
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Oxytocin: Each participant will self-administer 40 IU intranasal Oxytocin (OT)
  Oxytocin: 40 IU oxytocin nasal spray
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 100 | 100
score on a scale | 0.90 (0.12) | 1.21 (0.12)

2. Primary Outcome: Laboratory Intimate Partner Aggression Intensity (IPA)
Description: Intensity of laboratory-based IPA was assessed using the Taylor Aggression Paradigm (TAP). IPA intensity is operationalized as the volume of "shock" administered on a 1-10 (1 is least intense, 10 is most intense) scale using the computer based paradigm in response to "losing" trials.
  TAP is a fictitious reaction time competition among partners. Participants are told that a winning trial required them to deliver a shock to their partner that ranged from 1 to 10 intensity for a duration of their choosing. A losing trial resulted in them receiving a shock from their partner (administered through two electrodes attached to the index and middle fingers of the nondominant hand). In reality, all participants received an identical sequence of "winning" or "losing" trials (and corresponding shocks) generated by the TAP software. IPA was operationalized as the average intensity (volume) and duration of shocks administered in response to "losing" trials.
Time Frame: 10 minutes from start to end of TAP
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 100 | 100
units on a scale | 4.8 (2.2) | 4.3 (2.0)

3. Primary Outcome: Laboratory Intimate Partner Aggression (IPA) Duration
Description: Laboratory IPA Duration was measured by the length of time participants administered "shocks" in the Taylor Aggression Paradigm (TAP). Measured in milliseconds. Greater number of milliseconds represents a longer shock.
  TAP is a fictitious reaction time competition among partners. Participants are told that a winning trial required them to deliver a shock to their partner that ranged from 1 to 10 intensity for a duration of their choosing. A losing trial resulted in them receiving a shock from their partner (administered through two electrodes attached to the index and middle fingers of the nondominant hand). In reality, all participants received an identical sequence of "winning" or "losing" trials (and corresponding shocks) generated by the TAP software. IPA was operationalized as the average intensity (volume) and duration of shocks administered in response to "losing" trials.
Time Frame: 10 minutes from start to end of TAP
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 100 | 100
milliseconds | 405.5 (113.2) | 414.4 (117.0)

4. Secondary Outcome: Change in Cortisol
Description: Change in salivary cortisol measured between Time 4 (before the laboratory aggression paradigm) and Time 5 (after the laboratory aggression paradigm).
  Participants completed the VAS at 8 timepoints:
  Minute 0 (pre-OT/placebo) (Time 1) Minute 5 (pre-OT/placebo) (Time 2) OT/placebo administered at minute 10 Minute 40 (Time 3) Minute 45 - alcohol cue paradigm began Time 4 (immediately after alcohol cue) Minute 65 - TAP began Time 5 (immediately after TAP began) Time 6 (15 minutes after TAP) Time 7 (30 minutes after TAP) Time 8 (60 minutes after TAP)
  Higher salivary cortisol is indicative of higher stress response and lower salivary cortisol is indicative of lower stress response.
Time Frame: Measured between Time 4 (before the laboratory aggression paradigm) and Time 5 (after the laboratory aggression paradigm).
Measure: Mean (95% Confidence Interval); unit: ul/dL
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 100 | 100
ul/dL | 0.11 [0.09 to 0.13] | 0.11 [0.09 to 0.12]

5. Secondary Outcome: Change in Subjective Aggression
Description: Mean change in subjective aggression scores as measured by a Visual Analogue Scale (VAS) between time point 4 (after alcohol cue) and 5 (during Taylor Aggression Paradigm, TAP).
  Participants completed the VAS at 8 timepoints:
  Minute 0 (pre-OT/placebo) (Time 1) Minute 5 (pre-OT/placebo) (Time 2) OT/placebo administered at minute 10 Minute 40 (Time 3) Minute 45 - alcohol cue paradigm began Time 4 (immediately after alcohol cue) Minute 65 - TAP began Time 5 (immediately after TAP began) Time 6 (15 minutes after TAP) Time 7 (30 minutes after TAP) Time 8 (60 minutes after TAP)
  This 100mm Visual Analogue Scale (VAS) was anchored on a Likert-type scale from 0 (not at all/no aggression) to 10 (extremely/maximum aggression). The scale is set to 100mm in length, and the lowest value is a 0 (zero), representing no aggression and and highest value is a 10 (ten) representing extreme aggression.
Time Frame: Change is aggression measured between time point 4 (after the alcohol cue) and 5 (during Taylor Aggression Paradigm).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 100 | 100
score on a scale | 0.31 (0.10) | 0.41 (0.09)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Oxytocin | Control
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 6/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=100) | Control (N=100)
Lightheadedness (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Upper Respiratory Infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Nosebleed
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) — 1- car accident 1 - finger laceration
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — planned procedure

LIMITATIONS AND CAVEATS:
Ability to estimate anticipated power was limited by absence of prior studies examining effects of OT on aggression using TAP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT03046836/Prot_SAP_002.pdf
  • Informed Consent Form (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT03046836/ICF_001.pdf